IRB Pro00081972 Version 11/06/17

## **Data Analyses and Statistical Considerations**

We will perform descriptive analyses to determine engagement and feasibility. Linear mixed modeling will be used to test for across group differences in DASH adherence and other secondary outcomes. Our model will include group, time, and a group by time interaction, and will be fitted with a full maximum likelihood method using all data. As this is a feasibility study, we have estimated sample size from our previous text messaging trial where we saw strong engagement; 50% texted daily and 85% texted at least 2 days/week.